CLINICAL TRIAL: NCT06895941
Title: Predictive Value of PET/CT for Efficacy of Neoadjuvant Immunotherapy in Non-small Cell Lung Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Unable to support implementation.
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chang Chen, Chief Physician, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: PETici
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer (NSCLC); Neoadjuvant Immunotherapy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Diagnostic Test: PET — Exploring the predictive value of PET/CT metabolic parameters for the efficacy of neoadjuvant immunotherapy in non-small cell lung cancer.

SUMMARY:
The aim of this study was to investigate the enhancement of FAPI PET/CT metabolic parameters in predicting the efficacy performance of neoadjuvant immunotherapy using the pCR status of surgically resected specimens of lung cancer as the gold standard.

ELIGIBILITY:
Inclusion Criteria:(1) aged 18 years or older; (2) pathological diagnosis of non-small cell lung cancer; (3) lesions resectable by surgery; (4) no EGFR mutation or ALK mutation; (5) eligible for indications of neoadjuvant immunotherapy for lung cancer.

-

Exclusion Criteria:(1) patients who had used any other antitumor drugs or radiotherapy; (2) comorbidities with other malignant neoplastic diseases or severe cardiovascular diseases; (3) uncontrollable diabetes mellitus or fasting blood glucose level higher than 11 mmol/L on the test day; (4) pregnancy or recent pregnancy plan; (5) distant metastasis.

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer patients receiving neoadjuvant immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
FAPI PET/CT predicts efficacy | 2025.3.1-2027.3.1
  AUC predicted by FAPI PET/CT for neoadjuvant immunotherapy in lung cancer.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No